CLINICAL TRIAL: NCT02074189
Title: Adjuvant Chemotherapy Following Radical Cystectomy to Treat Locally Advanced Bladder Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Zhiwen Chen, M.D,Ph.D, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012XLC02-1; 2012XLC02 (Other Grant/Funding Number: 2012XLC02,Third Military Medical University,China)
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant Chemotherapy (Active Comparator): Adjuvant Chemotherapy(Gemcitabine, Cisplatin):Gemcitabine 1000 mg/m2 iv,D1,D8,D15;cisplatin 70 mg/m2 iv,D2.With 4 cycles. Treatment begins between 1-5 weeks after radical operation (within 42 days is recommended)
  Interventions: Drug: Gemcitabine, Cisplatin
- Control (No Intervention): No immediate post-surgery treatment. Patients undergo observation followed by cisplatin and gemcitabine as in arm I at local relapse, or receive intravenously chemotherapy with cisplatin and gemcitabine at multiple metastases

INTERVENTIONS:
Drug: Gemcitabine, Cisplatin — Gemcitabine 1000 mg/m2 iv,D1,D8,D15;cisplatin 70 mg/m2 iv,D2.With 4 cycles. Treatment begins between 1-5 weeks after radical operation (within 42 days is recommended)
  Other Names: GCT
  Arms: Adjuvant Chemotherapy

SUMMARY:
Effect of adjuvant chemotherapy to control tumor progression in patients after cystectomy for locally advanced bladder cancer.

DETAILED DESCRIPTION:
Effect of adjuvant chemotherapy based on Gemcitabine and Cisplatin to control tumor progression in patients after cystectomy for locally advanced bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older, estimated life expectancy ≥ 6 months.
2. Pathologically confirmed localized invasive bladder cancer following standardize radical cystectomy and pelvic lymphadenectomy.
3. Transitional cell carcinoma of bladder, stage pT3N0M0.Transitional cell carcinoma may be with or without squamous cell carcinoma and/or adenocarcinoma components.
4. Electrocorticography(ECOG) performance status 0-2.
5. Blood routine:Absolute neutrophil count (ANC) ≥ 1500/μL,White blood cell count ≥ 3000/μLPlatelets ≥ 100,000/μL,Hemoglobin ≥ 10.0 g/dL,
6. Total serum bilirubin≤ 1.5 x upper limit of normal (ULN).Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase(SGOT)) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase (SGPT)) ≤ 2.5 x upper limit of normal (ULN).
7. Creatinine clearance rate,Ccr ≥ 60%
8. ECG：no arrhythmias, no myocardial infarction.

   * Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
   * Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests,and other study procedures.

Exclusion Criteria:

1. Past history of systemic chemotherapy
2. Serious heart and lung dysfunction.
3. Associated with central or peripheral neuropathy greater than 2 grade.
4. Evidence of distant metastasis beyond the pelvis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-03; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
cancer progressive free survival rate | 60 months

SECONDARY OUTCOMES:
overall survival | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwen Chen, M.D,Ph.D, Principal Investigator — Southwest Hospital, China
Locations (1):
- Southwest hospital,China, Chongqing, Chongqing Municipality, China